CLINICAL TRIAL: NCT03793920
Title: Behavioral Exploration of Cognitive and Emotional Alterations in Adult Individuals Exposed to Alcohol During the Prenatal Period
Brief Title: Effects of Prenatal Alcohol Exposure on Emotional and Cognitive Abilities in Adults
Acronym: ALTEMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015_76; 2017-A00843-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-12-18; First posted 2019-01-04 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Prenatal Alcohol Exposure
Keywords: Prenatal alcohol exposure; Emotional; Cognition; Addiction; Fetal Alcohol Syndrome
MeSH Terms: conditions — Behavior, Addictive; Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PEA patients without alcohol disorder (Experimental): A group of 36 PEA patient without alcohol-dependence (AD), performing 6 behavioral tasks.
  Interventions: Other: Facial Emotion Test
- PEA patients with alcohol disorder (Sham Comparator): A group of 36 PEA participants, currently alcohol-dependent, performing 6 behavioral tasks.
  Interventions: Other: Facial Emotion Test
- Healthy controls with AD father (Sham Comparator): A group of 36 non-alcohol-dependent controls whose father was alcohol-dependent during their childhood and adolescence, performing 6 behavioral tasks.
  Interventions: Other: Facial Emotion Test
- Healthy controls without AD father (Sham Comparator): A group of 36 non-alcohol-dependent controls whose father was not alcohol-dependent during their childhood and adolescence, performing 6 behavioral tasks.
  Interventions: Other: Facial Emotion Test

INTERVENTIONS:
Other: Facial Emotion Test — All tasks will be delivered using a laptop and E-Prime 2 software (Psychology Software Tools, Inc., Pittsburgh), which will also be used to collect behavioral responses.

SUMMARY:
Hypothesis:

Individuals presenting with prenatal alcohol exposure (PEA) show emotional abilities deficits, and imbalance between the two systems involved in decision-making according to dual-process models, namely an under-activated reflective system (involved in deliberate behaviors) and an over-activated affective-automatic one (involved in impulsive behaviors).

Primary objective:

To explore performance (as a percentage of correct answers) in an emotional facial expression decoding task in PEA participants compared to controls without alcohol disorder.

DETAILED DESCRIPTION:
Each participant will undergo 2 visits :

First visit :

* Checking inclusion and non-inclusion criteria
* Note of information and consent form
* Record of concomitant treatments and anamnestic elements
* Alcohol, Tobacco, and Toxic Consumption
* Urinary Toxicity Test for Control Groups
* Laterality test (Hecaen, 1984)
* Brief visual and auditory acuity test
* Standardized psychiatric interview (Mini International Neuropsychiatric Interview - MINI)

Second visit = Experimental testing

* State-Trait Anxiety Inventory, Beck Depression Inventory, Inventory of Interpersonal Problems, Toronto Alexithymia Scale (TAS-20).
* Participant installation and testing: 6 behavioral tasks on a computer (also used to collect responses, except for task 2, see details below) :

Task 1 (MAIN): Test for recognition of facial emotions Task 2: 'Reading the Mind in the Eyes Test' (Decoding of complex emotional states) Task 3: Emotional evaluation of natural scenes Task 4: Target detection (measure of attentional bias towards alcohol-related stimuli) Task 5: Go / No-Go evaluating the interactions between inhibition processes and auto-affective system Task 6: "N-back" evaluating the interactions between working memory and automatic-affective system

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged between 18 and 60 years
* Able to understand and to speak French
* Able to understand Note of information and to sign consent form
* Available health insurance
* Normal (or corrected to normal) vision and audition
* For women: Negative pregnancy test or menopausal for at least one year
* For Group 1 only : PEA criteria and no alcohol consumption within the three days preceding the experiment.
* For Group 2 only : PEA criteria, diagnosed with severe alcohol addiction and currently abstinent (for at least 15 days).
* For Group 3 only : Non-alcohol-dependent controls. No alcohol consumption within the three days preceding the experiment and father diagnosed with severe alcohol addiction.
* For Group 4 only : Non-alcohol-dependent controls. No alcohol consumption within the three days preceding the experiment.

Exclusion Criteria:

* Refusal of participation after clear and fair information on the study.
* Visual or auditory sensory disability to participate in the study.
* Benzodiazepines and / or Antipsychotic concomitant treatment.
* History of (or current) neurologic disease
* History of (or current) psychiatric disorder (apart alcohol-dependence for the PEA-alcohol-dependent group)
* Psychoactive Substance Use or Abuse other than tobacco and alcohol.
* Pregnant or breast-feeding women.
* Underage (<18 yo) or adults under guardianship, judicial protection, or deprived of liberty.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-11-08 (Actual); Primary Completion 2022-11-11 (Estimated); Study Completion 2022-11-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of correct answers of an emotional facial expression (EFE) | one day
  Performance of an emotional facial expression (EFE) decoding task in EPA subjects and compare it to non-alcohol dependent controls

SECONDARY OUTCOMES:
Psychopathological assessment by Mini International Neuropsychiatric Interview MINI | one day
  Presence of psychiatric disorders by a standardized psychiatric interview
Percentage of correct answers ant latency of behavioral answers | one day
  Performance of behavioral tasks
State-Trait-Anxiety Inventory (STAI) score | one day
  Score at STAI STAI is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis
Beck Depression Inventory score | one day
  Score at Beck Depression Inventory The BDI consisted of twenty-one questions about how the subject has been feeling in the last week. Each question had a set of at least four possible responses, ranging in intensity. (0) I do not feel sad/ (1) I feel sad./ (2) I am sad all the time and I can't snap out of it/ (3) I am so sad or unhappy that I can't stand it.
  When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-off scores were as follows:0-9: indicates minimal depression/ 10-18: indicates mild depression/ 19-29: indicates moderate depression/ 30-63: indicates severe depression.
Toronto Alexithymia Scale TAS-20 score | one day
  Score at TAS-20 The Toronto Alexithymia Scale is a measure of deficiency in understanding, processing, or describing emotions. The current version has twenty statements rated on a five-point Likert scale. ( range : Strongly disagree/Disagree/ Neither agree nor disagree/ Agree/ Strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier COTTENCIN, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - CSAPA, Lille
  - CHRU Lille, Fontan2, Lille